CLINICAL TRIAL: NCT07055087
Title: A Randomized, Double-blind, Placebo-controlled, 104-week Proof-of-concept Study to Evaluate the Efficacy of Intravenous Prasinezumab in Participants With Parkinson's Disease Carrying a Severe Mutation in the GBA Gene
Brief Title: Prevent Cognitive Decline in GBA-associated Parkinson's Disease
Acronym: PreCoDe
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PreCoDe; 2024-513496-40-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-03; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-05

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Cognitive function; GBA; anti-α-synuclein; monoclonal antibody
MeSH Terms: conditions — Parkinson Disease | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prasinezumab (Experimental): prasinezumab 1500 mg monthly infusion
  Interventions: Drug: Prasinezumab
- Sodium chloride 0,9% infusion (Placebo Comparator): saline infusion (0,9 % sodium chloride) monthly infusion
  Interventions: Drug: Sodium Chloride

INTERVENTIONS:
Drug: Prasinezumab — Prasinezumab 1500 mg monthly infusion
  Arms: Prasinezumab
Drug: Sodium Chloride — Saline infusion (0,9 % sodium chloride) monthly infusion
  Arms: Sodium chloride 0,9% infusion

SUMMARY:
This is a proof-of-concept trial to investigate the efficacy of prasinezumab to slow or prevent cognitive decline in people with Parkinson's disease carrying a severe mutation in the GBA (glucocerebrosidase) gene. The duration of the intervention per patient will be 104 weeks with monthly infusions. The investigators plan to enroll 120 participants (60 participants per treatment arm). This study will be conducted across Europe in the following countries: France, Germany, Italy, Luxembourg, Spain, Sweden, UK.

DETAILED DESCRIPTION:
This is a proof-of-concept (POC) prospective, multicenter, randomized, double-blind, placebo-controlled clinical trial to investigate the efficacy of the intravenously (IV) applied monoclonal anti-α-synuclein antibody prasinezumab to slow or prevent cognitive decline in people with Parkinson's disease (PD) carrying a severe mutation in the GBA (glucocerebrosidase) gene (PDGBA_severe). The duration of the intervention per patient will be 104 weeks with monthly infusions. The investigators plan to enroll 120 participants (60 participants per treatment arm).

This study will be conducted across Europe in the following countries: France, Germany, Italy, Luxembourg, Spain, Sweden, UK.

Randomization will be 1:1 prasinezumab (1500mg) versus placebo (saline infusion). Randomization will be stratified by sex, age group (< 55 years vs ≥ 55 years), and baseline Montreal Cognitive Assessment (MoCA) (≤ 25) to ensure balance of these factors between the prasinezumab and placebo group.

Participants, aged 35 to 80 years, diagnosed with PD and carrying a known severe mutation in the GBA gene according to the definition for PD (see Supplemental Table 1 for a list of applicable mutations). MoCA at Screening must be ≥ 21.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of PD according to MDS-Criteria.
2. Known heterozygous severe GBA mutation (based on PD-related pathogenicity).

   --> In case of slow recruitment after 6 months, inclusion of the GBA risk variant E326K as back-up strategy is possible (based on PD-related pathogenicity). This will be communicated by the sponsor beforehand.
3. MoCA ≥ 21.
4. HY in dopaminergic ON ≤3.
5. 35 to 80 years of age at the time of signing the Informed Consent.
6. Able and willing to provide written informed consent and to comply with the study protocol according to the International Council for Harmonization (ICH) and local regulations.

Exclusion Criteria:

Current or Past Medical History:

1. Known pathogenic mutation carriers of the following familial PD genes: PRKN, PINK1, DJ1, LRRK2.
2. Medical history indicating a Parkinsonian syndrome other than sporadic PD (progressive supranuclear palsy, multiple system atrophy, drug-induced parkinsonism, essential tremor, primary dystonia).
3. A diagnosis of a significant CNS disease other than PD.
4. Previous, current or planned (within next 2 years) treatment with Deep Brain Stimulation (DBS) or ablation with high-intensity focused ultrasound or planned treatment with these within the next 2 years.
5. History of brain MRI scan indicative of clinically significant abnormality of prior hemorrhage or ischemic infarction > 1 cm3, > 3 lacunar infarctions, vascular encephalopathy with white matter lesions according to Fazekas grade III. Clinical routine brain MRI scan must be available within 2 years before Screening.
6. Concomitant disease or condition, or treatment thereof that could interfere with the conduct of the study, or that would, in the opinion of the Investigator, pose an unacceptable risk to the participant in this study or interfere with the participant's ability to comply with study procedures or abide by study restrictions, or with the ability to interpret safety data, including:

   1. Autoimmune disease (however, well controlled conditions such as quiescent rheumatoid arthritis [RAS], controlled type I diabetes, or mild-to-moderate psoriasis not requiring systemic medications may be acceptable after discussion with Sponsor).
   2. History of malignancy within 5 years prior to screening, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, non-metastatic prostate cancer, or Stage I uterine cancer.
   3. Any active infectious disease at Screening.
   4. Current, or history of, alcohol or drug abuse or other dependence (except nicotine dependence) within one year before Screening. Drug and/or alcohol abuse within 12 months prior to screening, in the investigator's judgment (except nicotine dependence, Marijuana use is not allowed [this includes all forms of cannabidiol and tetrahydrocannabinol even if given for therapeutic use]).
   5. Any febrile illness within one week prior to first dose administration.
   6. Any current psychiatric diagnosis according to Diagnostic and Statistical Manual of Mental Disorders fifth edition (DSM-5), International Statistical Classification of Diseases and Related Health Problems 10th Revision (ICD-10) or equivalent, that may interfere with the participant's ability to perform the study and all assessments (e.g., major depression (BDI-II >28, mental retardation, schizophrenia, bipolar disorder, etc.).

      Note: Mild depression, depressive mood or mild anxiety arising in the context of PD, are not exclusionary.
   7. Acute suicidality, as evidenced by a) Question 5 ("Lifetime"/"Since last visit") on the Columbia- Suicide Severity Rating Scale (C-SSRS), indicating active suicidal ideation with any intent to act, at Screening or baseline (Day 1), or answering "yes" for Question 3 ("In the Past Month"/"Since last visit") on the C-SSRS, indicating active suicidal ideation with any methods (not plan) without intent to act, at Screening or baseline (Day 1)
7. The following cardiovascular conditions:

   1. Myocardial infarction in the last 12 months prior to baseline.
   2. Known history or documentation of uncontrolled bradycardia on more than one occasion within three months prior to baseline.
   3. Resting pulse rate (PR) greater than 110.
   4. Known history or documentation of uncontrolled hypertension on more than one occasion within three months prior to baseline.
   5. Clinically significant cardiovascular disease including any of the following: unstable angina, decompensated congestive heart failure, clinically significant arrhythmias.
8. Clinically significant abnormalities in laboratory test results at the Screening visit, including hepatic and renal panels, complete blood count, and urinalysis, including:

   1. Total bilirubin, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 times the upper limit of normal (ULN).
   2. Serum creatinine > 1.5 times the ULN.
   3. Hematocrit (Hct) less than 35% for males and less than 32% for females, or absolute neutrophil cell count of < 1500/μL (with the exception of a documented history of a chronic benign neutropenia), or platelet cell count of < 100,000/μL; international normalized ratio (INR) > 1.4
   4. A clinically significant abnormal thyroid-stimulating hormone (TSH) test.
   5. A positive urine drug screen for a drug of abuse. For participants treated with selegiline, the amphetamine drug abuse test should be based on the results from a urine assay by liquid chromatography-mass spectrometry which is able to differentiate false positives from true positives for methamphetamine. For participants treated with benzodiazepines: A positive urine drug screen for benzodiazepines is allowed, provided that the prescription has been on a stable dosage for 90 days prior to baseline.
   6. Positive result for acute or chronic infectious hepatitis B virus (HBV; [i.e., hepatitis B surface antigen (HBsAg positive test)]), for hepatitis C virus (HCV), or HIV 1 or 2. Successfully treated patients with HCV (undetectable HCV RNA) are eligible for enrollment. Participants who are immune due to HBV natural infection or HBV vaccination are eligible.
9. Female participants of childbearing potential without highly effective contraceptive methods (that result in a failure rate of < 1% per year) during the treatment period and for at least 90 days (or longer if required by local regulations) after the last dose of study drug.

   1. A female participant is considered to be of childbearing potential if she is post-menarchal, has not reached a post-menopausal state (> 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (i.e. removal of ovaries, fallopian tubes, and/or uterus).
   2. Examples of highly effective contraceptive methods (with a failure rate of < 1% per year) include bilateral tubal ligation, vasectomized partner, established, proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
   3. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the participant. Periodic abstinence (e.g., calendar, ovulation or post ovulation methods) and withdrawal are not acceptable methods of contraception.
10. Lactating or pregnant female participants. Female participants of childbearing potential must have a negative serum pregnancy test result during screening prior to initiation of study drug.

    Medications and treatments:
11. If on treatment with symptomatic therapy: no stable dosage for at least 90 days before Baseline of following drugs/drug classes:

    1. dopamine agonists,
    2. MAO-B inhibitors,
    3. COMT inhibitors,
    4. amantadine, and/or
    5. levodopa. Note: pumps for continuous levodopa treatment are acceptable if on stable dosage for at least 90 days before Baseline
12. Manifest Gaucher's Disease and treatment for Gaucher's Disease:

    1. enzyme replacement therapy (ERT),
    2. substrate reduction therapy (SRT). Note: A second PD-associated risk variant in the GBA gene, namely E326K and T396M is allowed
13. Anti-epileptic medication for non-seizure-related treatment which has not remained on a stable dosage for at least 90 days prior to baseline and not planned to remain stable during the study.
14. Anti-depressant or anxiolytic use that has not remained on a stable dosage for at least 90 days prior to baseline and not planned to remain stable during the study.
15. Use of any of the following medications within 90 days prior to baseline: typical neuroleptics, metoclopramide, flunarizine, amoxapine, amphetamine derivatives, reserpine, mazindol, methamphetamine, methylphenidate, norephedrine, phentermine, phenylpropanolamine, modafinil, alpha methyldopa, cocaine.

    Note: Amantadine, quetiapine, and clozapine are allowed but should be on a stable dose for at least 90 days prior to baseline.
16. Prior and concomitant participation in a putative disease-modifying investigational trial with surgical, or stem cell intervention in PD.
17. Prior and concomitant participation in an investigational clinical trial with symptomatic or disease modifying PD treatment within 90 days (or 5 half-lives of the drug, whichever is longer) before baseline.
18. Any prior treatment with an investigational PD-related vaccine (including active immunization or passive immunotherapy with monoclonal antibodies).
19. Prior participation in any prasinezumab study or study with other compounds targeting alpha-synuclein.
20. Receipt of any non-PD investigational product or device, or participation in a non-PD drug research study within a period of 90 days (or 5 half-lives of the drug, whichever is longer) before baseline.
21. Receipt of any monoclonal antibody or investigational immunomodulator within 180 days (or 5 half-lives, whichever is longer) before baseline (e.g., monoclonal antibodies, intravenous immunoglobulin [IVIG], interleukin 2 [IL-2], interleukin 12 [IL-12], interferon or immunosuppressive drugs).
22. Immunomodulating drugs including oral corticosteroids within 90 days prior to baseline.
23. Allergy to any of the components of prasinezumab such as citrate, trehalose and polysorbate (Tween) 20 or a known hypersensitivity or an IRR to the administration of any other monoclonal antibody.

    Note: Enrollment in a non-interventional study may be allowed if approved in advance by the Sponsor.

    Procedural:
24. Any contraindications to obtaining a brain MRI (if brain MRI was not already performed within 2 years before of Screening, see exclusion criteria) (e.g., claustrophobia unresponsive to reassurance or low dose of an anxiolytic agent, tooth implants).
25. Donation of blood over 500 mL within three months prior to Screening.
26. For participants consenting to provide optional CSF samples by lumbar puncture (LP): LP will only be performed if the participant does not have any contraindication to undergoing an LP including: INR > 1.4 or other coagulopathy, platelet cell count of < 120,000/μL, infection at the desired LP site, taking anti-coagulant medication within 10 days of baseline (Note: low dose aspirin [acetylsalicylic acid and clopidogrel is permitted], severe degenerative arthritis of the lumbar spine, suspected non-communicating hydrocephalus or intracranial mass, prior history of spinal mass or trauma is/are identified. Participants failing to meet these criteria can still participate in the study and all other study assessments (with the exception of LP) as appropriate.

    Regulatory & Administrational:
27. Patients under legal supervision or guardianship.
28. Participants who are not fluent in the national language.
29. Residing in a nursing home or assisted care facility.
30. Participating in any other interventional clinical trial.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2031-05 (Estimated)

PRIMARY OUTCOMES:
Parkinson's Disease Cognitive Composite Score (PDCCS) | week 104
  To assess the efficacy of prasinezumab compared with placebo on cognitive function at week 104 measured by the Parkinson's Disease Cognitive Composite Score (PDCCS).
  Composite score that includes the following cognitive tests:
  * LNS (Attention)
  * Derived-Sem. Fluency-Animal T-Score (Executive function)
  * Derived-Delayed Recall T-Score (Memory)
  * MoCA (Global cognition) Per single Test: Group Mean and Standard Deviation (SD) at Baseline = reference ZBaseline = (xBaseline - Group MeanBaseline) / SDBaseline ZFollow-up = (xFollow-up - Group MeanBaseline) / SDBaseline
  Mean of Z-Scores of relevant Tests per Patient per Visit Min-Max: n.a. (higher values mean a better outcome)

SECONDARY OUTCOMES:
Cognitive function (MoCA_z) | week 104
  Cognitive function measured by MoCA_z (Montreal Cognitive Assessment demographically-corrected z-value) Min-Max: 0 - 30 (higher values mean a better outcome)
PD-MCI | week 104
  Percentage of participants with diagnosis of PD-MCI defined by MDS Level II criteria
PDD | week 104
  Percentage of participants with diagnosis of PDD
MDS-UPDRS I-IV | week 104
  International Parkinson and Movement Disorder Society (MDS) Unified Parkinson's Disease Rating Scale (UPDRS) part I-IV Min-Max: 0 - 272 (lower values mean a better outcome)
Levodopa-equivalent dosage | week 104
  Levodopa-equivalent dosage [mg]
Cognitive function per cognitive domain: Attention and working Memory (1/2) | week 104
  Cognitive function per cognitive domain: Attention and working Memory: Trail Making Test Part A (TMT A) Min-Max: 0 - 100 seconds (lower values mean a better outcome)
Cognitive function per cognitive domain: Attention and working Memory (2/2) | week 104
  Cognitive function per cognitive domain: Attention and working Memory: Wechsler Adult Intelligence Scale (WAIS) IV: Letter-Number Span (LNS) Min-Max: 0 - 21 (higher values mean a better outcome)
Cognitive function per cognitive domain: executive (1/3) | week 104
  Cognitive function per cognitive domain: Executive: Verbal Fluency (animal fluency) Score: number of named animals (higher values mean a better outcome)
Cognitive function per cognitive domain: executive (2/3) | week 104
  Cognitive function per cognitive domain: Executive: Stroop interference Min-Max: 0 - n.a. (lower values mean a better outcome)
Cognitive function per cognitive domain: executive (3/3) | week 104
  Cognitive function per cognitive domain: Executive: Trail Making Test (TMT) part B Min-Max: 0 - 300 seconds (lower values mean a better outcome)
Cognitive function per cognitive domain: memory (1/2) | week 104
  Cognitive function per cognitive domain : Memory: Hopkins verbal learning test (HVLT) Delayed Recall Min-Max: 0-12 (higher values mean a better outcome)
Cognitive function per cognitive domain: memory (2/2) | week 104
  Cognitive function per cognitive domain : Memory: Wechsler Memory Scale (WMS) IV: logical memory I Min-Max: 0 - 50 (higher values mean a better outcome)
Cognitive function per cognitive domain: visuospatial (1/2) | week 104
  Cognitive function per cognitive domain: Visuospatial: Benton's Judgment of Line Orientation Min-Max: 0 - 30 (higher values mean a better outcome)
Cognitive function per cognitive domain: visuospatial (2/2) | week 104
  Cognitive function per cognitive domain: Visuospatial: Hooper Visual Organization Test Min-Max: 0 - 30 (higher values mean a better outcome)
Cognitive function per cognitive domain: language (1/2) | week 104
  Cognitive function per cognitive domain: Language: Boston naming Min-Max: 0 - 60 (higher values mean a better outcome)
Cognitive function per cognitive domain: language (2/2) | week 104
  Cognitive function per cognitive domain: Language: Wechsler Adult Intelligence Scale (WAIS) IV: similarities Min-Max: 0 - 33 (higher values mean a better outcome)

OTHER OUTCOMES:
Exploratory: cognitive function (MoCA_z) | week 104
  Cognitive function measured by PDCCS in the prasinezumab and placebo group separately compared to MoCA_z values (Montreal Cognitive Assessment demographically-corrected z-value) PDCCS is a composite score (see primary endpoint for details)
Exploratory: Cognitive function (MoCA ≥ 26) | week 104
  Cognitive function measured by PDCCS in the prasinezumab versus placebo group in participants who were cognitively normal at baseline as defined by MoCA ≥ 26.
  PDCCS is a composite score (see primary endpoint for details)
Exploratory: Cognitive function (PD-MCI) | week 104
  Cognitive function measured by PDCCS in the prasinezumab versus placebo group in participants who had PD-MCI at baseline as defined by MoCA ≤ 25.
  PDCCS is a composite score (see primary endpoint for details)
Exploratory: IADL | week 104
  Cognitive-driven Instrumental Activities of Daily Living (IADL) as measured by the FAQ (Functional Activities Questionnaire) cognitive score provided by the patient and caregiver separately.
  Min-Max: 0-30 (lower values mean a better outcome)
Exploratory: cognitive IADL impairment | week 104
  Percentage of participants with more cognitive than motor IADL impairment defined by FAQ quotient > 1.008.
  Min-Max: 0 - 100 %
Exploratory: PDQ-39 | week 104
  Quality of life as measured by PDQ-39 (Parkinson's Disease Quality of Life Questionnaire).
Exploratory: MCI, RBD, orthostatic hypotension | week 104
  Percentage of participants with either (or combined) MCI, REM-sleep-behaviour disorder (RBD; assessed by RBD questionnaire) and orthostatic hypotension (assessed by Schellong test).
Exploratory: NPI-Q | week 104
  Percentage of hallucinations as assessed by NPI-Q (Neuropsychiatric Inventory questionnaire) Min-Max: 10 - 120 (lower values mean a better outcome)
Safety outcome measures | from first dose administration up to 12 weeks after cessation of treatment
  Number of patients with abnormal laboratory values.
Safety outcome measures | from first dose administration up to 12 weeks after cessation of treatment
  Number of patients with AEs
Safety outcome measures | from first dose administration up to 12 weeks after cessation of treatment
  Number of patients with ADAs
Safety outcome measures | from first dose administration up to 12 weeks after cessation of treatment
  Number of patients with treatment-emergent abnormal laboratory values and abnormal laboratory values reported as AEs
Safety outcome measures | from first dose administration up to 12 weeks after cessation of treatment
  Number of patients with abnormal ECG assessments
Safety outcome measures | from first dose administration up to 12 weeks after cessation of treatment
  Number of patients with abnormal blood pressure [systolic and diastolic]
Safety outcome measures | from first dose administration up to 12 weeks after cessation of treatment
  Number of patients with abnormal heart rate and orthostatic changes.
Safety outcome measures | from first dose administration up to 12 weeks after cessation of treatment
  Number of patients with exacerbation of motor and psychiatric side-effects (including C-SSRS).
Exploratory: biomarkers serum/CSF | week 104
  Quantitative measures and prevalence of pathological profiles of biomarkers:
  α-synuclein seeding activity (yes/no)
Exploratory: biomarkers serum/CSF | week 104
  Quantitative measures and prevalence of pathological profiles of biomarkers:
  α-synuclein seeding activity LAG [hours] Min-Max: 0 - 40 (higher values mean better outcome)
Exploratory: biomarkers serum/CSF | week 104
  Quantitative measures and prevalence of pathological profiles of biomarkers:
  α-synuclein seeding activity iMAX [no unit] Min-Max: 0 - 100 (lower values mean better outcome)
Exploratory: biomarkers serum/CSF | week 104
  Quantitative measures and prevalence of pathological profiles of biomarkers:
  α-synuclein seeding activity AUC [no unit] Min-Max: 0 - 1000 (lower values mean better outcome)
Exploratory: biomarkers serum/CSF | week 104
  Quantitative measures and prevalence of pathological profiles of biomarkers: Glucosphingolipids panel (lower values mean better outcome)
Exploratory: biomarkers serum/CSF | week 104
  Quantitative measures and prevalence of pathological profiles of biomarkers: Neurofilament-light chain [pg/ml] Min-Max: 0 - 10.000 (lower values mean better outcome)
Exploratory: biomarkers serum/CSF | week 104
  Quantitative measures and prevalence of pathological profiles of biomarkers: Abeta_42 [pg/ml] Min-Max: 0 - 2.000 (higher values mean better outcome)
Exploratory: biomarkers serum/CSF | week 104
  Quantitative measures and prevalence of pathological profiles of biomarkers: Abeta_40 [pg/ml] Min-Max: 0 - 10.000 (lower values mean better outcome)
Exploratory: biomarkers serum/CSF | week 104
  Quantitative measures and prevalence of pathological profiles of biomarkers: total-Tau [pg/ml] Min-Max: 0 - 10.000 (lower values mean better outcome)
Exploratory: biomarkers serum/CSF | week 104
  Quantitative measures and prevalence of pathological profiles of biomarkers: phospho-Tau [pg/ml] Min-Max: 0 - 200 (lower values mean better outcome)
Exploratory: biomarkers serum/CSF | week 104
  Quantitative measures and prevalence of pathological profiles of biomarkers: inflammation panel in plasma and/or serum and if applicable in CSF [no unit] (lower values mean better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Kathrin Brockmann, Prof. Dr., Principal Investigator — University Hospital Tuebingen
Locations (8):
- Sorbonne University, Pitié-Salpêtrière Hospital, Paris, France
- University Hospital Tubingen, Tübingen, Germany
- Italy (2):
  - University of Brescia and ASST Spedali Civili of Brescia, Brescia
  - Fondazione IRCCS Ca' Granda Policlinico Hospital, Milan
- University of Luxemburg, Luxembourg, Luxembourg
- Hospital Universitario HM Puerta del Sur, Madrid, Madrid, Spain
- Karolinska University of Stockholm, Stockholm, Sweden
- University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided